CLINICAL TRIAL: NCT03043443
Title: Melatonin for Alcohol Use Disorder Patients With Sleeping Problems
Brief Title: Melatonin Use for Sleep Problems in Alcohol Dependent Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Bernard Le Foll, Dr., Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 099-2016
Record Dates: First submitted 2017-02-01; First posted 2017-02-06 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Alcohol-Related Disorders
Keywords: sleep; Alcohol dependence; Melatonin
MeSH Terms: conditions — Alcohol-Related Disorders; Alcoholism | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Subjects with Alcohol use disorder and sleep problems will be recruited and assigned randomly to the active treatment Melatonin or Placebo arms.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): participants will receive placebo 1 capsule/day 1 hour before sleeping for 4 weeks
  Interventions: Drug: Placebo
- Melatonin (Active Comparator): participants will receive melatonin 1 capsule (5mg)/day 1 hour before sleeping for 4 weeks
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — Natural health product for sleep problems treatment
  Other Names: melatonin 5 mg oral tablets
  Arms: Melatonin
Drug: Placebo — Lactose containing pills
  Other Names: Lactose pills
  Arms: Placebo

SUMMARY:
A double blind Randomized Controlled Trial with two arms will be used. Subjects with Alcohol use disorder and sleep problems will be recruited and assigned randomly to the active treatment Melatonin or Placebo arms. All subjects will be assessed at baseline for demographics. Sleeping problems will be the primary outcome of the study, and it will be measured by the Pittsburgh sleep quality index (PSQI) scale.

DETAILED DESCRIPTION:
A double blind Randomized Controlled Trial with two arms will be used. Subjects with Alcohol use disorder and sleep problems will be recruited and assigned randomly to either Melatonin or Placebo arms. All subjects will complete some forms on the REDCap system such as contact information list, concomitant medication, Time Line Follow Back (TLFB), Fagerstrom test for nicotine dependence (FTND), Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI), AUD criteria, and Alcohol use disorder identification test (AUDIT). Sleeping problems will be the primary outcome of the study, and it will be measured by the Pittsburgh sleep quality index (PSQI) scale where score 5 or more indicated a sleeping problem. Women in child-bearing period will be asked to do a urine pregnancy test to exclude pregnancy. After verifying eligibility, the participants will come to pick up the medication (Melatonin or placebo) blister together with a sleep hygiene document and will start taking the medication for 4 weeks. All subjects will then be followed-up at the end of 1 month of treatment and PSQI score will be measured. This step will be completed either online by sending an email link through or the participants can come to a personal visit to complete the second PSQI form. Also, this last visit/email will contain side effects questionnaire, TLFB, BDI, BAI. All the participants will be required to bring/send back the medication blister pack to do a pill count and check all the missing pills.

ELIGIBILITY:
Inclusion Criteria:

* Age: 19 or older
* AUD in any stage
* Sleep problems in the past month
* PSQI score > 5 at baseline
* Participants must agree not to use other sleep aid during the study
* Women capable of becoming pregnant must agree to use contraceptives during study

Exclusion Criteria:

* Pregnancy, lactation or plans to become pregnant during the study timeline.
* Use of other sleep aid in the past month (either prescribed or over the counter remedies)
* Use of benzodiazepines and/or Z- drugs: (zaleplon, zolpidem and zopiclone) in the past month
* Known allergy to melatonin
* Participants taking immunosuppressive drugs.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
PSQI score | 1 month
  The primary outcome of the study is PSQI score. This will be analyzed by the difference in the global score before and after the use of melatonin versus placebo. Score > 5 indicates a sleep problem.

SECONDARY OUTCOMES:
PSQI subscales | 1 month
  Secondary outcome measures will include the subscales of PSQI: 1) subjective quality of sleep; 2) sleep onset latency; 3) sleep duration; 4) sleep efficiency; 5) presence of sleep disturbances; and 6) presence of daytime disturbances, as an indication of daytime alertness.
  As according to previous studies, melatonin showed a significant decrease in sleep onset latency and an improvement in daytime alertness.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard LeFoll, MD, Principal Investigator — Centre of addiction and mental health
Locations (2):
- Canada (2):
  - Centre for Addiction and Mental Health, Toronto, Ontario
  - Center for Addiction and Mental Health, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No